CLINICAL TRIAL: NCT07331376
Title: Improving Perceived Stress, Anxiety, and Sleep Quality Among Nursing Students: Enhancing Resilience Through Emotional Freedom Techniques
Brief Title: EFT and Resilience in Nursing Students
Acronym: Emotional
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Leyla SEZGİN, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07.11.2025-218893
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Emotional Well-being; Sleep Quality; Nursing Students
Keywords: Nursing Students; Sleep Quality; Emotional Freedom Techniques (EFT)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The sample for this study consisted of individuals who volunteered to participate in the research from among the students enrolled in the Nursing Department of the Faculty of Health Sciences at Muş Alparslan University during the 2025-2026 academic year.
  Simple random sampling was used to select the sample for the study. Students who met the participation criteria and agreed to participate in the study were randomly assigned to the experimental and control groups from among all students in the population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Freedom Techniques (EFT) Intervention Group (Experimental): This arm applies Emotional Freedom Techniques (EFT) to nursing students to reduce stress- and anxiety-related sleep disturbances and to improve sleep quality, duration, and restorative function.
  Participants receive EFT sessions twice weekly for 8 weeks (45 minutes per session) conducted by a certified EFT trainer or a qualified mental health nurse in a quiet, well-ventilated classroom or counseling room.
  Each session follows a structured sequence:
  Opening and awareness (grounding): Participants describe their current emotional and sleep-related state.
  SUDS assessment (pre-test): Participants rate discomfort levels regarding sleep difficulty on a 0-10 scale.
  EFT tapping sequence: Guided, sleep-focused tapping targeting stress, anxiety, and sleep concerns.
  Reflection and closing: Participants discuss emotional changes and relaxation effects post-intervention.
  The EFT intervention is designed to enhance psychological resilience, promote emotional regulation, and improve overall sl
  Interventions: Behavioral: Emotional Freedom Techniques
- Sham Emotional Freedom Techniques (Active Placebo Control Group) (Placebo Comparator): This arm involves an active placebo (sham) intervention designed to control for the non-specific effects of Emotional Freedom Techniques (EFT) such as attention, touch, and expectation of benefit.
  The procedure mimics the structure and appearance of genuine EFT sessions but omits its core therapeutic components-specifically, tapping on energy meridian points and the use of emotionally focused affirmations. The goal is to provide a credible comparison condition that elicits similar expectations of stress and sleep improvement while lacking the specific EFT mechanisms.
  Intervention Details:
  Purpose: To simulate the general relaxation and expectancy effects of EFT without including its specific active therapeutic elements.
  Total Duration: 8 weeks Session Frequency: 2 sessions per week Session Length: Approximately 45 minutes per session Setting: Quiet, comfortable classroom or consultation room Practitioner: Same instructor as in the genuine EFT group to maintain consistency
  Interventions: Other: PLESEBO
- Objectives of the Control Group (No Intervention): Isolating the Effect of the Intervention The control group helps determine whether observed improvements in perceived stress, anxiety, and sleep quality result specifically from the EFT intervention, rather than from external factors such as the passage of time, habituation, or natural recovery.
  Distinguishing the Placebo Effect In psychosocial and behavioral interventions, non-specific factors-such as receiving attention from a practitioner, participating in a structured activity, and the psychological expectation of improvement ("I will get better")-can independently produce beneficial outcomes.
  The control group is used to account for and measure these placebo-related effects.Demonstrating the Natural Process In the absence of an active therapeutic intervention, the control group allows observation of how perceived stress, anxiety levels, and sleep quality naturally fluctuate or change over time.

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques — Emotional Freedom Techniques
  Arms: Emotional Freedom Techniques (EFT) Intervention Group
Other: PLESEBO — PLESEBO
  Arms: Sham Emotional Freedom Techniques (Active Placebo Control Group)

SUMMARY:
The purpose of this study is to determine the effect of Emotional Freedom Technique (EFT) application on stress, anxiety, and sleep quality in nursing students.

The nursing education process can cause high levels of psychological and physiological stress in students due to many factors such as a heavy theoretical knowledge load, clinical practice stress, exam anxiety, and shift work. This situation results in increased anxiety and impaired sleep quality, thereby negatively affecting students' academic performance, clinical skills, and overall well-being.

In this context, the study aims to evaluate whether EFT, as a complementary method, is effective in reducing stress and anxiety levels in nursing students, as well as improving sleep quality.

It is believed that the results of this research will contribute to the development of alternative approaches that support psychological well-being in nursing education and will provide evidence-based data on the integration of EFT into educational programs.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of Emotional Freedom Technique (EFT) application on stress, anxiety, and sleep quality in nursing students.

The nursing education process can cause high levels of psychological and physiological stress in students due to many factors such as a heavy theoretical knowledge load, clinical practice stress, exam anxiety, and shift work. This situation results in increased anxiety and impaired sleep quality, thereby negatively affecting students' academic performance, clinical skills, and overall well-being.

In this context, the study aims to evaluate whether EFT, as a complementary method, is effective in reducing stress and anxiety levels in nursing students, as well as improving sleep quality.

It is believed that the results of this research will contribute to the development of alternative approaches that support psychological well-being in nursing education and will provide evidence-based data on the integration of EFT into educational programs.

Existing studies on EFT applications for nursing students show promising results in reducing exam/academic anxiety and general stress levels; for example, some pre-post and small controlled studies have reported decreases in both stress and exam anxiety (Patterson, 2016; Vural, 2019). However, these studies have limitations such as sample size, use of comparison groups, and lack of long-term follow-up; therefore, the number of RCT (randomized controlled trial) studies with strong methodological design in the nursing student population is still limited.

Sleep quality is a strong determinant of both cognitive functioning and mood in students; when stress and anxiety levels are impaired, sleep quality can deteriorate, and conversely, improved sleep can contribute to a reduction in psychological symptoms. Studies investigating the direct effect of EFT on sleep quality are also increasing: studies conducted in various age groups and clinical populations report that EFT can improve sleep parameters or provide subjective sleep quality improvement, while some studies report mixed effect sizes or heterogeneous results in group comparisons (Souilm et al., 2022; Kalroozi et al., 2022; Özcan, 2025).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the Nursing Department at Muş Alparslan University,
* Be 18 years of age or older,
* Agree to participate in the study voluntarily,
* Have no psychiatric diagnosis or regular use of psychotropic medication.

Exclusion Criteria:

Students who do not regularly participate in the application process,

* Students who do not complete the data collection forms in full,
* Students who report physical or psychological discomfort during the EFT application process.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Levels from Baseline to Week 8 Measured by the Perceived Stress Scale (PSS) | UP TO 8 WEEKS
  Baseline and Week 8 (after completion of intervention)

SECONDARY OUTCOMES:
Change in Subjective Sleep Duration from Baseline to Week 8 as Reported by Participants | UP TO 8 WEEKS
  Baseline and Week 8 (after completion of intervention)

IPD SHARING:
Plan to Share IPD: No